CLINICAL TRIAL: NCT00063817
Title: Renal Allograft Tolerance Through Mixed Chimerism (ITN010ST)
Brief Title: Reducing the Risk of Transplant Rejection: Simultaneous Kidney and Bone Marrow Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN010ST; DAIT NKD03 (Other: Immune Tolerance Network)
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: End-stage Renal Disease; Renal Transplantation; Kidney Transplantation
Keywords: End-stage renal disease; Renal Transplant; Bone Marrow Transplant; nonmyeloablative conditioning regimen
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation Conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditioning Regimen (Experimental): Cyclophosphamide intravenously (IV) on days -5 and -4 with respect to transplantation; MEDI-507 on days -1, 0, and 1 (after a test dose of 0.1 mg per kg on day -2); and cyclosporine A IV and thymic irradiation on day -1. Hemodialysis was performed before and 14 hours after each dose of cyclophosphamide.Kidney transplantation was followed by IV infusion of donor bone marrow. Oral cyclosporine A was administered daily postoperatively, with target trough blood levels of 250 to 350 ng per milliliter; the dose was tapered and discontinued over a period of several months.
  Amendment applicable to the 4th and 5th participant: rituximab on days -7 and -2; and prednisone, 2 mg per kg per day starting on the day of transplantation with tapering over the next 10 days.
  Interventions: Drug: Conditioning Regimen

INTERVENTIONS:
Drug: Conditioning Regimen — Cyclophosphamide 60 mg per kilogram (kg) of body weight per day intravenously (IV) on days -5 and -4 with respect to transplantation; humanized anti-CD2 monoclonal antibody (MEDI-507) 0.6 mg per kg on days -1, 0, and 1 (after test dose of 0.1 mg per kg on day -2); and cyclosporine A 5 mg per kg IV and thymic irradiation (700 cGy) on day -1. Hemodialysis was performed before and 14 hours after each dose of cyclophosphamide.Kidney transplantation was followed by IV infusion of donor bone marrow. Oral cyclosporine A was administered postoperatively, 8 to 12 mg per kg per day, with target trough blood levels of 250 to 350 ng per milliliter; the dose was tapered and discontinued over a period of several months. Protocol amendment that applied to participant 4 and 5: rituximab, 375 mg per square meter of body-surface area days -7 and -2; and prednisone, 2 mg per kg per day starting on the day of transplantation with tapering over the next 10 days.
  Other Names: nonmyeloablative preparative regimen

SUMMARY:
This study will examine the safety and effectiveness of a combination kidney and bone marrow transplant from a relative with the same (or nearly the same) blood cell type as the transplant recipient. An investigational medication will be given prior to and after the transplant to help protect the transplanted kidney from attack by the body's immune system.

DETAILED DESCRIPTION:
Of the two currently available treatments for kidney failure, long-term dialysis and kidney transplantation, only kidney transplantation provides a potential cure. After a kidney transplant, the body's immune system recognizes the kidney as foreign and tries to attack and destroy it in a process called rejection. To avoid rejection, participants must take medications called immunosuppressants or anti-rejection drugs. It is believed that by transplanting bone marrow at the same time as a solid organ such as a kidney, a state of "mixed chimerism" (a mixing of the donor and recipient's immune system) can be achieved. Mixed chimerism may prevent rejection without the need for anti-rejection drugs.

Participants in this study will receive a simultaneous bone marrow and kidney transplant from the same living related donor in an attempt to establish mixed chimerism. Prior to transplantation, participants will undergo a "conditioning regimen" involving cyclophosphamide chemotherapy, radiation to the thymus gland, and four immunosuppressive medications: cyclosporine A, a man-made antibody known as rituximab to suppress B cells, a short course of steroids, and a T-cell depleting antibody known as MEDI-507. MEDI-507 is an investigational medication that has not been approved by the FDA. The primary goal of the study is to investigate the safety of the conditioning regimen and its ability to promote mixed chimerism so that the transplanted kidney is not destroyed. The study will also determine whether participants with mixed chimerism can eventually be safely removed from long-term immunosuppressive therapy following transplantation.

Participants will be assessed before and after transplantation and will be followed ≤36 months.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease (ESRD) without prior sensitization (defined as Panel Reactive Antibody [PRA] greater than 20%) within the 60 days prior to transplant as measured by cytotoxicity assays, ELISA, and flow cytometry;
* Undergoing a first or second transplant;
* Receiving a transplant from a living related donor who is ABO (blood type) compatible and haploidentical (3, 4, or 5 antigen match by serologic typing);
* Cardiac ejection fraction greater than 40%;
* Forced expiratory volume (FEV1) greater than 50%;
* Liver function tests, bilirubin, and coagulation studies less than 2 X normal;
* White blood cells greater than 2000/mm^3; abd
* Platelets greater than 100,000/mm^3

Exclusion Criteria:

* Positive donor lymphocyte cross-match;
* HIV-1 infected;
* Positive hepatitis B surface antigen (HbsAg);
* Hepatitis C virus infected;
* History of cancer;
* Prior dose-limiting radiation therapy;
* Pregnant, breastfeeding, or planning pregnancy within the time frame of the study;
* Enrolled in another investigational drug study within 30 days prior to study entry; or
* Receiving maintenance immunosuppression within 3 months before the conditioning regimen begins

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2003-06; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Graft Survival Twenty-Four Months Post Transplantation | 24 months (2 Years) Post Transplantation
  Defined by kidney transplant survival at month 24 post transplantation with successful withdrawal of cyclosporine following transplantation, in the absence of maintenance immunosuppression.

SECONDARY OUTCOMES:
Participant Survival | Up to thirty-six months (3 Years) Post Transplantation
  During the three-year post-transplant follow-up period for enrolled participants.
Graft Survival | Up to thirty-six months (3 Years) Post Transplantation
  During the three-year post-transplant follow-up period for enrolled participants.
Change from Baseline in Renal Function Using Serum Creatinine | Up to thirty-six months (3 Years) Post Transplantation
  Changes in serum creatinine levels from baseline through post transplantation follow-up period.
Number of Episodes of Acute or Chronic Graft Versus Host Disease (GVHD) | From Week 1 through thirty-six months (3 Years) Post Transplantation
  Evaluations for suspected GVHD, including biopsies as appropriate, during routine and/or for cause assessments.
Number of Adverse Events | Participant enrollment through <=thirty-six months (3 Years) Post Transplantation
  As defined by protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David H. Sachs, MD, Principal Investigator — Department of Medicine, Massachusetts General Hospital; A. Benedict Cosimi, MD, Principal Investigator — Department of Medicine, Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Kawai T, Cosimi AB, Spitzer TR, Tolkoff-Rubin N, Suthanthiran M, Saidman SL, Shaffer J, Preffer FI, Ding R, Sharma V, Fishman JA, Dey B, Ko DS, Hertl M, Goes NB, Wong W, Williams WW Jr, Colvin RB, Sykes M, Sachs DH. HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2008 Jan 24;358(4):353-61. doi: 10.1056/NEJMoa071074. PMID 18216355
- See also: National Institute of Allergy and Infectious Diseases website — https://www.niaid.nih.gov/
- See also: Click here for the Immune Tolerance Network website — http://www.immunetolerance.org